CLINICAL TRIAL: NCT03453801
Title: The Role of CD4+ Memory Phenotype, Memory, and Effector T Cells in Vaccination and Infection Adaptive Immune Responses and Repertoire in Influenza Vaccination and Infection
Brief Title: The Role of CD4+ Memory Phenotype, Memory, and Effector T Cells in Vaccination and Infection
Acronym: SLVP030
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Grant, Assistant Professor of Medicine (Infectious Diseases), Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-31256; U19AI057229-11 (NIH)
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Influenza; Healthy
Keywords: Inactivated, influenza vaccine quadrivalent; Live, attenuated influenza vaccine quadrivalent; Young children; Identical twins
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MZ twins 2-5 yo (Experimental): Monozygotic twins, 2-5 yo (annual return): In 2014-2015, individual twin participants will be given FluMist® a live, attenuated influenza vaccine quadrivalent (LAIV4) intranasally. Vaccine non-naive participants will return annually for flu immunization and for blood samples on Days 0, 7 and 60 post-immunization. Vaccine naive children will receive two immunizations in the first year, 28 days apart then return annually for flu immunization. Blood samples will be obtained on Days 0, 7 and 60 post second-immunization. Beginning in 2015-2016, participants in this arm will receive Fluzone® inactivated influenza vaccine quadrivalent (IIV4) as an intramuscular (IM) injection annually following Advisory Committee on Immunization Practices (ACIP) recommendation against LAIV4.
  Interventions: Biological: Fluzone®; Biological: FluMist®
- Non-twins 6 mo-10 yo (Experimental): Non-twins 6 mo-10 years (annual return): In 2014-2015, participants between 6-23 mo will be given Fluzone® inactivated influenza vaccine quadrivalent (IIV4) IM then switch to FluMist® a live, attenuated influenza vaccine quadrivalent (LAIV4) intranasally starting at age 24 months in annual follow-up. Participants aged 24 mo-8 yo will be given LAIV4 at enrollment and for annual follow-up. However, if LAIV4 is contraindicated, the child will continue with IIV4. Participants 9-10 yo will be given IIV4 annually. Vaccine non-naive participants will return annually for flu immunization and for blood samples on Days 0 and 60 post immunization. Vaccine naive children will get two doses of vaccine the first year then return annually for flu immunization and blood samples on Day 0 and 60 post second immunization. Beginning in 2015-2016, all participants in this arm will receive Fluzone® inactivated influenza vaccine quadrivalent (IIV4) annually following ACIP recommendation against LAIV4.
  Interventions: Biological: Fluzone®; Biological: FluMist®
- Non-twins 6-12 mo Flu/MMRV Naïve (Experimental): Non-twins 6-12 mo Flu/MMRV Naïve (annual return): In 2014-2015, participants 6-12 mo who are flu and MMRV naïve will be given Fluzone® inactivated influenza vaccine quadrivalent (IIV4) as an IM injection. In Year 1, participants will return for a second flu immunization at least 28 days later and for blood samples on Days 0 and 60 post-second immunization and on Day 60 post MMRV (to be given by primary care physician). In Years 2-5, participants will return annually for Fluzone® IIV4 flu immunization and for blood samples on Days 0 and 60 post-immunization.
  Interventions: Biological: Fluzone®

INTERVENTIONS:
Biological: Fluzone® — Fluzone® Quadrivalent (IIV4; inactivated influenza virus vaccine): The pediatric dose (6-35 months) will be supplied in a prefilled, single dose syringe, 0.25 mL (no preservative). Each 0.5 mL dose of Fluzone® Quadrivalent (36 months-adult) will be supplied in a prefilled, single dose syringe, 0.5 mL (no preservative). Both formulations given IM.
  Other Names: IIV4
Biological: FluMist® — FluMist® Quadrivalent: live, attenuated influenza virus vaccine quadrivalent, given by intranasal spray
  Other Names: LAIV4
  Arms: MZ twins 2-5 yo; Non-twins 6 mo-10 yo

SUMMARY:
The purpose of this study is provide a better understanding of the adaptive immune response to the licensed influenza vaccines in children.

DETAILED DESCRIPTION:
This is a Phase I study of up to 100 healthy children, ages 6 months to 10 years of age, who will receive either Flumist® live, attenuated influenza virus vaccine, quadrivalent (LAIV4) or the current Fluzone® inactivated influenza vaccine, quadrivalent (IIV4). The volunteers will be enrolled into one of 3 Groups. Volunteers will return each year until 2018-2019 for annual flu immunizations and study visits. Questionnaires will be administered annually to record demographic characteristics, vaccination history, exposure to animals, day care and medically attended illness. There are no exclusions for gender, ethnicity or race.

Volunteers in the Non-twin Flu/MMRV naive group will also receive the measles, mumps, rubella and varicella (MMRV) vaccine at approximately 12-15 months of age (to be administered by the volunteers' personal pediatrician, not as a study vaccine). They will then come for a study visit to collect blood 60 days later.

Each twin is counted as a single participant. All reporting numbers reflect the number of participants, not the number of twin pairs.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy non-twins 6 months - 10 years old, or 2-5 year old identical (MZ) twins.
2. Willing to complete the informed consent process (including assent for minors 7 years old and above).
3. Availability for follow-up for the planned duration of the study - annually until 2018-2019 influenza vaccination season
4. Acceptable medical history by review of inclusion/exclusion criteria and vital signs.
5. Non-twin flu/MMRV naive group: Willing to have primary care physician immunize child with the MMRV vaccine and return for a study visit approximately 60 days later.

Exclusion Criteria:

1. Prior off-study vaccination with the current year's seasonal influenza vaccine.
2. Life-threatening reactions to previous influenza vaccinations
3. Allergy to egg or egg products, or to vaccine components
4. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
5. History of immunodeficiency (including HIV infection)
6. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
7. Chronic Hepatitis B or C.
8. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible in all groups; inhaled steroid use is not permissible)
9. Malignancy
10. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
11. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
12. Receipt of blood or blood products within the past 6 months or planned used during the study.
13. Receipt of Inactivated vaccine 14 days prior to study enrollment, or planned vaccinations prior to completion of last study visit ( ~ 28 Day after study vaccination)
14. Receipt of live, attenuated vaccine within 60 days prior to enrollment of planned vaccination prior to completion of last study visit (~ 28 Day after study vaccination)
15. Need for allergy immunization (that cannot be postponed) during the study period.
16. History of Guillain-Barré syndrome
17. Use of investigational agents within 30 days prior to enrollment or planned use during the study.
18. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or planned donation prior to completion of the last visit.
19. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Frequency of antigen-specific T memory phenotype cells (TMP) | Day 0 to Day 60
  The percentage of cells with the various antigen-specific T memory phenotypes will be determined.

SECONDARY OUTCOMES:
T cell receptor (TCR) repertoire analysis deep phenotyping by mass cytometry (CyTOF) | Day 0 to Day 60
  The TCR repertoire encompasses the different sub-types of T-cell receptors of the immune system.
Deep phenotyping by mass cytometry (CyTOF) | Day 0 to Day 60
  Deep phenotyping is the analysis of phenotypic abnormalities of the individual components of the phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L Dekker, MD, Principal Investigator — Stanford University; Mark M Davis, PhD, Principal Investigator — Stanford University; Philip M Grant, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No